# 临床研究受试者知情同意书

方案名称:索凡替尼联合卡瑞利珠单抗及mFOLFOX6方案二线治疗晚期胰腺癌的探索性临床研究

方案版本号: V2.3, 2023年12月12日

知情同意书版本号: V2.4, 2023年12月12日

研究机构: 中山大学肿瘤防治中心

主要研究者: 骆卉妍

您将被邀请参加一项临床研究。本知情同意书提供给您一些信息以帮助您决定是否参加 此项临床研究。请您仔细阅读,如有任何疑问请向负责该项研究的研究者提出。

您参加本项研究是自愿的。本次研究已通过本研究机构伦理审查委员会审查。

### 【研究概述】

告知研究基本信息,包括:参加研究的总人数,研究持续时间,受试者参加研究的预期持续时间。本研究是一项单臂、单中心 II 期临床研究,计划入组 37 例受试者。本研究预计入组时间为 2023 年 9 月至 2025 年 9 月。预计研究结束时间为 2026 年 9 月。

### 【研究目的】

初步评价索凡替尼联合卡瑞利珠单抗及 mF0LF0X6方案二线治疗晚期胰腺癌是否有生存 获益,为晚期胰腺癌二线及后线治疗探讨可行性策略。

胰腺癌被称为癌中之王,是预后最差的常见实体恶性肿瘤之一,具有恶性程度高、预后差的特点,全球总体发病率和死亡率逐年上升,2020年导致全球 46.6万例死亡,居所有恶性肿瘤第七位。我国胰腺癌死亡率居所有恶性肿瘤第六位,在 2020年新发病例达 12.5万例,死亡病例达 12.2万例。经预测,至2030年胰腺癌将成为全球第二大癌症死因。 胰腺癌主要治疗手段包括手术切除、化疗、放疗和生物治疗等,但治疗效果均不理想,是治疗效果最差的恶性肿瘤之一。5年总生存率(0S)不到 10%,在恶性肿瘤中最低,预测 2030年,胰腺癌死亡率将仅次于肺癌。目前手术治疗结合辅助治疗仍然是胰腺癌患者能获得长期生

存机会的唯一方法,然而 80%以上的晚期胰腺癌患者丧失了手术的可能,积极的行内科治疗 尤为重要。局部进展期或合并远处转移的胰腺癌总体治疗效果不佳,中位生存期在 6-9 个 月,建议开展相关临床研究。

2022 年 CSCO 指南推荐转移性胰腺癌患者一线治疗方案,应根据患者体能状态进行选择,对于体能状态良好的患者,可以考虑联合方案,体能状态较差患者选择单药化疗(GEM 或替吉奥单药)或最佳支持治疗。目前对于转移性胰腺癌的治疗仍以化疗为主。对于已经失去手术机会且 KPS≥70 分的转移性胰腺癌患者,标准治疗一般采取联合化疗。其中,一线化疗方案目前有 2 个国际公认标准:奥沙利铂+伊立替康+5-FU/亚叶酸(FOLFIRINOX)三药方案和白蛋白紫杉醇+吉西 他滨(AG)两药方案,其中 FOLFIRINOX 方案预期有效率为 30%,预期生存 11-12 个月,AG 方案预期有效率为 25%~30%,预期生存 8.5-11 个月。AG 方案和 FOLFIRINOX方案可以互为一线二线,即患者一线耐药后可以更换另一种方案继续治疗,对两种方案的回顾性研究显示,使用顺序不影响患者预后。尽管白蛋白结合紫杉醇联合吉西他滨或 FOLFIRINOX 化疗方案已被证明对胰腺癌患者有显著的生存获益,但其进一步的疗效仍存在挑战。

二线治疗方案目前 CSCO 指南推荐体能状态良好的患者接受纳米脂质体伊利替康联合 5-FU/LV; NAPOLI-1 研究为随机对照III期临床研究,纳米脂质体伊立替康+5-FU/LV 的 mOS 为 6.1 个月,5-FU/LV 为 4.2 个月(HR=0.67, P=0.012),两组差异有统计学意义。NAPOLI-1 研究共纳入亚洲患者 132 例(韩国和中国台湾),亚洲患者的亚组分析结果显示,纳米脂质体伊立替康+5-FU/LV 的 mOS 为 8.9 个月,5-FU/LV 为 3.7 个月(HR = 0.51, P = 0.025)。其他推荐方案还包括:一线使用吉西他滨为基础的方案,二线建议以 5-FU 为基础的方案;一线使用 5-FU 类为基础的方案,二线建议使用吉西他滨为基础的方案;对于术后发生远处

转移者,若距离辅助治疗结束时间>6个月,除选择原方案全身化疗外,也可选择替代性化疗方案;参加临床研究。

mFOLFOX6方案为氟尿嘧啶和奥沙利铂为基础的化疗方案,不同的用药剂量和顺序已被证明氟尿嘧啶和奥沙利铂为基础的化疗方案三线治疗转移性胰腺癌的有效性。其中 CONKO-003研究中,OFF 方案的 OS(5.9 个月 vs 3.3 个月)和 PFS(2.9 个月 vs 2.0 个月)都高于 FF 方案。Yoo C 等开展的研究中证实,mFOLFOX6 方案的 ORR(7% vs 0)和主要研究终点 6 个月的 PFS 率(30% vs 27%) 略高于 mFOLFIRI.3 外,OS 和 PFS 均不及 mFOLFIRI.3 方案。此外,SEQUOIA 研究还对 Pegilodecakin(PEG)联合 FOLFOX 与 FOLFOX 方案的疗效进行了对比, 结果显示联合治疗组和单纯化疗组疗效相当。

综上,目前针对晚期胰腺癌二线治疗,单一的治疗手段疗效欠佳,免疫联合治疗也未满足晚期胰腺癌患者的治疗需求,仍需探索新的治疗方法。

#### 【研究过程】

在进入筛选期之前,您需要阅读本知情同意书,如果您充分了解了本知情同意书的内容, 并且自愿参与本项研究,您需要签署本知情同意书。接下来您需要在医院接受以下检查和评估,这些检查是您常规医疗检查的一部分,即使您不参加本次研究,也可能需要做这些检查, 来帮助您的医生为您选择合适的治疗方案。在完成了这些检查和评估后,如果您不符合入组 要求,您的研究医生将与您讨论其他的治疗选择。

- 核对入选/排除标准;
- 记录人口学数据;
- 既往病史、既往用药和合并用药;
- 不良事件记录:
- 身高、体重、生命体征(体温,脉搏,呼吸频率,血压);
- ECOG 评分:

- 体格检查: 一般情况,头面部,皮肤,淋巴结,眼(巩膜、瞳孔),耳部,鼻部,咽喉部,口腔、呼吸系统,心血管系统,腹部(包含肝脾),生殖-泌尿系统,肌肉骨骼,神经系统,精神状况;(注:试验期间须进行全面的体格检查,只需记录异常情况,如与筛选期相比无变化,则不需重复记录);
- 实验室检查: 血常规, 血生化, 尿常规, 大便常规, 凝血功能, 甲状腺功能, 血HCG 检测(有潜在生育能力的受试者); HBV, HCV, HIV 检查; • 十二导联心电图;
  - 心脏超声检查;
- 影像学评估:胸部+腹部+盆腔 CT 增强扫描。如存在造影剂过敏等其他原因不 能耐受增强扫描受试者,应采用MRI 检查;

在完成了所有这些评价和检查之后,您也许无法满足所有入组条件而不能参加本研究,但还有其它的替代疗法来治疗您的疾病,包括其它的药物或对症治疗。您的研究医生将和您讨论其他最佳治疗选择。

### 【研究治疗】

化疗方案及用法用量:

- 索凡替尼: 索凡替尼推荐日剂量为 250mg, 每日一次, 连续给药:
- 卡瑞利珠单抗: 给药剂量固定为 200mg, 在联合用药期间每 14 天给药一次, 维持治疗期间每 21 天给药一次, 用药最多满 2 年后停药;
- 化疗方案 (mFOLFOX6, 奥沙利铂+亚叶酸钙+氟脲嘧啶): 奥沙利铂 85mg/m2 d1+CF 400mg/m2 d1+5-FU 400mg/m2 d1/2400mg/m2 持续静注 (civ) 46h, 每 14 天给药一次, 共 8-12 个周期, 具体周期数由研究者综合判断。

### 【参加研究可能的风险和不适】

和其他治疗肿瘤类的药物一样,接受索凡替尼和卡瑞利珠单抗治疗可能出现一 些不良事件,包括但不局限于下列各项。

(1) 索凡替尼主要不良反应如下:索凡替尼的安全性数据来自 8 项单药治疗的临床研究,总计 718 例晚期肿瘤患者接受起始剂量 ≥300 mg,每日 1 次,连续服药的用药方案;其中 357 例患者来自 2 项在神经内分泌瘤患者中进行的关键性 III

期随机双盲对照研究[1 项为非胰腺来源的神经内分泌瘤研究(SANET-ep),含 193 例接受索凡替尼的患者;另 1 项为胰腺神经内分泌瘤研究(SANET-p),含 164 例接受索凡替尼的患者]。在 718 例患者中,发生率≥20% 不良反应包括:蛋白尿、高血压、血胆红素升高、腹泻、血白蛋白降低、血甘油三酯升高、血促甲状腺激素升高、疲乏 / 乏力、腹痛、外周水肿、血尿酸升高、出血。

按系统器官分类、首选术语和发生频率汇总的索凡替尼在 8 项研究的 718 例患者中的不良反应见下表。发生频率分为:十分常见( $\geq$ 10%),常见(1%  $\sim$  10%,含 1%),偶见(0.1% $\sim$ 1%,含 0.1%),罕见(0.01% $\sim$ 0.1%,含 0.01%),十分罕见(<0.01%)。在每个发生频率分组内,不良反应按发生率从高至低依次列出:

| 肾脏及泌尿系统疾病 | |
|------------|--------------------------|
| 十分常见 | 蛋白尿 |
| 血管及淋巴管类疾病 | |
| 十分常见 | 高血压、出血 |
| 偶见 | 高血压危象 |
| 胃肠系统疾病 | |
| 十分常见 | 腹泻、腹痛、便秘 |
| 全身性疾病及给药部位 | 立各种反应 |
| 十分常见 | 疲乏/乏力、外周水肿 |
| 内分泌系统疾病 | |
| 十分常见 | 甲状腺功能减退症 |
| 各类神经系统疾病 | |
| 十分常见 | 头痛 |
| 各种肌肉骨骼及结缔组 | 且织疾病 |
| 常见 | 关节痛 |
| 心脏器官疾病 | |
| 常见 | 常见 窦性心动过缓 |
| 各类检查 | |
| 十分常见 | 血胆红素升高、血白蛋白降低、血甘油三酯升高、血促 |
| | 甲状腺激素升高、血尿酸升高、血小板计数降低、心电 |

| | 图 T 波或 ST-T 段异常、尿中带血、血钾降低、中性粒 |
|----|-------------------------------|
| | 细胞计数降低、血肌酐升高 |
| 常见 | 血钠降低、血红蛋白升高、血尿素升高、血糖降低 |

# (2) 卡瑞利珠单抗主要不良反应如下:

卡瑞利珠单抗在临床研究中以单药治疗或与化疗联合治疗中观察到的不良反应,并按照系统器官分类和发生频率列出这些不良反应。发生频率定义如下:十分常见(≥1/10),常见(≥1/100至<1/10),偶见(≥1/1,000至<1/10),罕见(≥1/10,000至<1/10),不良反应按发生率从高到低依次排列。

| | 单药治疗 | 与化疗联合治疗 |
|---|---|---|
| 感染和侵染 | | |
| 常见 | 肺部感染,上呼吸道感染 <sup>®</sup> | 肺部感染,尿路感染,上呼吸道感染 <sup>°</sup> |
| 偶见 | 皮肤软组织感染 <sup>b</sup> ,尿路感染 | 局部炎症 <sup>°</sup> |
| 罕见 | 脓毒性休克 | |
| 血液和淋巴系 | | |
| 十分常见 | 贫血,白细胞减少症 | 贫血,中性粒细胞减少症,白细胞减少症,血小板减少症,淋巴细胞减少症 |
| 常见 | 中性粒细胞减少症,血小板减少症,<br>淋巴细胞减少症 | 单核细胞减少症 |
| 偶见 | 淋巴结病 | 发热性中性粒细胞减少症 |
| 免疫系统疾病 | | |
| 常见 | 输液相关反应 <sup>d</sup> | 输液相关反应 <sup>d</sup> |
| 内分泌疾病 | | |
| 十分常见 | 甲状腺功能减退 | 甲状腺功能减退 |
| 常见 | 甲状腺功能检查异常 <sup>6</sup> ,甲状腺功能亢进 | 甲状腺功能检查异常。,甲状腺功能亢进 |
| 偶见 | 垂体激素检查异常 <sup>f</sup> ,肾上腺功能不<br>全,肾上腺皮质激素检查异常 <sup>g</sup> ,甲状<br>腺炎 | 垂体激素检查异常 <sup>f</sup> ,甲状腺炎,抗甲状腺抗体阳性,垂体炎,肾上腺皮质激素检查异常 <sup>g</sup> |
| 罕见 | 垂体炎 | |

| | 单药治疗 | 与化疗联合治疗 |
|---|---|---|
| 代谢和营养病组 | T<br>武 | |
| 十分常见 | | 食欲下降 <sup>h</sup> ,低蛋白血症 <sup>i</sup> |
| 常见 | 食欲下降 <sup>1</sup> ,低蛋白血症 <sup>1</sup> ,低钠血症,<br>高脂血症,低钾血症 | 高脂血症,低钾血症,糖尿病,低钠血症 |
| 偶见 | 低磷血症,糖尿病 | 低磷血症 |
| 精神病症 | | |
| 常见 | | 失眠 <sup>i</sup> ,嗜睡 |
| 偶见 | 失眠 <sup>i</sup> ,嗜睡,晕厥 | |
| 罕见 | 昏迷 | |
| 神经系统疾病 | | |
| 常见 | 头晕 | 头晕,感觉减退 <sup>k</sup> ,头痛 |
| 偶见 | 头痛,感觉减退 <sup>k</sup> ,肌无力综合征 <sup>1</sup> | 肌无力综合征¹,外周神经病变™,认知障碍 |
| 罕见 | 外周神经病变™,脑炎 | |
| 眼部疾病 | | |
| 常见 | | 干眼症,眼痛,流泪增加 |
| 偶见 | 结膜炎 | 结膜炎,视物模糊 |
| 罕见 | 干眼症,视物模糊,眼痛 | |
| 心血管疾病 | , | |
| 常见 | 高血压 | 高血压,心动过速 <sup>n</sup> |
| 偶见 | 心电图 QT 间期延长,血压降低,心<br>肌酶谱检查异常°,心律不齐°,心动<br>过速 <sup>n</sup> ,急性冠脉综合征,肝血管瘤,<br>心动过缓,心肌炎,静脉血栓,潮红 | 心律不齐 <sup>3</sup> ,心动过缓,心力衰竭,心电图 QT 间期延长,血压降低,肝血管瘤,静脉血栓 |
| 罕见 | 心肌梗死,血管破裂,血管病,雷诺<br>现象 | |
| 呼吸、胸部和组 | ,<br>从膈疾病 | |
| 常见 | 肺炎 <sup>°</sup> ,咳嗽,胸部不适 <sup>°</sup> ,呼吸困难,<br>鼻衄,咳痰 | 肺炎 <sup>°</sup> ,胸部不适 <sup>r</sup> ,胸腔积液 <sup>°</sup> ,咳嗽,鼻衄 |
| 偶见 | 咯血,呼吸衰竭,胸腔积液 <sup>3</sup> ,呼吸急促,发音困难,支气管炎,缺氧 | 咳痰,呼吸衰竭,呼吸急促 |

| | 单药治疗 | 与化疗联合治疗 |
|---|---|---|
| 罕见 | 哮喘 | |
| 胃肠道疾病 | | |
| 十分常见 | | 恶心, 便秘, 呕吐 |
| 常见 | 腹泻,恶心,腹痛 <sup>t</sup> ,呕吐,便秘,口<br>腔黏膜炎 <sup>t</sup> | 腹胀,腹泻,腹痛 <sup>¹</sup> ,呃逆,口腔黏膜炎 <sup>"</sup> ,<br>食管反流病,消化道出血 <sup>²</sup> ,牙龈牙周疾病<br>结直肠炎 <sup>*</sup> |
| 偶见 | 牙龈牙周疾病**,腹胀,口干,呃逆,结直肠炎*,口腔出血,消化道出血*,痔疮,不完全肠梗阻 | 口干,口腔出血,功能性胃肠紊乱 <sup>y</sup> ,口咽不适 <sup>z</sup> ,慢性胃炎 <sup>aa</sup> ,吞咽困难,消化道溃疡 <sup>bb</sup> |
| 罕见 | 功能性胃肠紊乱 <sup>x</sup> ,口腔扁平苔藓,口腔病,口咽不适 <sup>z</sup> ,马-魏二氏综合征(Mallory-Weiss syndrome),呕血,胃穿孔,胃食管反流病,吞咽困难,消化道溃疡 <sup>bb</sup> ,胰腺炎,食管瘘,慢性胃炎 <sup>aa</sup> ,异物感 | |
| 肝脏疾病 | | |
| 十分常见 | 天门冬氨酸氨基转移酶升高,丙氨酸<br>氨基转移酶升高、血胆红素升高 | 天门冬氨酸氨基转移酶升高,丙氨酸氨基转移酶升高,γ-谷氨酰转移酶升高,血胆红素<br>升高 |
| 常见 | γ-谷氨酰转移酶升高,血碱性磷酸酶<br>升高 | 血碱性磷酸酶升高 |
| 偶见 | 肝衰竭,药物诱导的肝损伤,免疫相<br>关性肝炎 | |
| 皮肤和皮下组织 | 只异常 | |
| 十分常见 | 反应性毛细血管增生症 | 反应性毛细血管增生症,皮疹 <sup>cc</sup> ,瘙痒 <sup>dd</sup> |
| 常见 | 皮疹 <sup>cc</sup> ,瘙痒 <sup>dd</sup> | 白癜风⁰ |
| 偶见 | 皮炎 <sup>ff</sup> ,白癜风 <sup>ee</sup> ,皮下出血 <sup>sg</sup> ,脱发,<br>掌跖红肿综合征,红斑 <sup>hh</sup> | 皮炎 <sup>ff</sup> ,脱发,红斑 <sup>bh</sup> ,银屑病,皮肤干燥 |
| 罕见 | 过敏性紫癜,毛细血管扩张症,银屑<br>病,皮肤肿块 | |
| 肌肉骨骼和结缔组织疾病 | | |
| 常见 | 肌肉骨骼疼痛 <sup>ii</sup> | 肌肉骨骼疼痛 <sup>ii</sup> |
| 偶见 | 关节炎 <sup>ij</sup> | 关节炎 <sup>ij</sup> |

| | 单药治疗 | 与化疗联合治疗 |
|---|---|---|
| 罕见 | 肌炎 | |
| 肾脏和泌尿系统 | 充疾病 | |
| 十分常见 | 蛋白尿 | 血肌酐升高 |
| 常见 | 血肌酐升高 | 蛋白尿 |
| 偶见 | 肾炎 <sup>kk</sup> | 肾炎 <sup>kk</sup> ,排尿困难,少尿 |
| 罕见 | 尿频 | |
| 全身性疾病及组 | 合药部位状况 | |
| 十分常见 | 乏力, 发热 | 乏力,水肿 <sup>11</sup> |
| 常见 | 水肿11,体重降低,体重增加 | 体重降低,发热,体重增加 |
| 偶见 | 寒战,流感样疾病,畏寒 | 疼痛"",休克 |
| 罕见 | 疼痛"",疲劳 | |
| 生殖系统及乳腺 | 泉疾病 | |
| 偶见 | 男性乳腺发育 | |
| 罕见 | 性功能障碍 | |
| 耳部疾病 | I | |
| 偶见 | 耳鸣 | 耳鸣 |
| 其他实验室检查 | | |
| 常见 | 脂肪酶升高,高尿酸血症,尿红细胞阳性,淀粉酶升高,大便潜血阳性,血糖升高,血乳酸脱氢酶升高,乙型肝炎 DNA 检测阳性 <sup>™</sup> | 高尿酸血症,其他实验室检查异常 <sup>60</sup> ,血糖升高,大便潜血阳性,血乳酸脱氢酶升高,凝血功能检查异常 <sup>60</sup> ,尿红细胞阳性,其他电解质紊乱 <sup>64</sup> ,其他尿常规检查异常 <sup>17</sup> |
| 偶见 | 其他电解质紊乱 <sup>99</sup> ,其他实验室检查异常 <sup>99</sup> ,其他心电图检查异常 <sup>95</sup> ,凝血功能检查异常 <sup>99</sup> ,其他尿常规检查异常 <sup>17</sup> | 淀粉酶升高,其他心电图检查异常 <sup>ss</sup> ,尿游离皮质醇降低 |

所示的不良反应频率可能不完全归因于卡瑞利珠单抗单药,也可能受潜在疾病或联合使用的其他药物影响。 以下术语代表描述某种病症的一组相关事件,而不是单一事件。发生频率参照涵盖的单一事件的最高发生率。

- a. 上呼吸道感染 (上呼吸道感染、鼻咽炎、喉部炎症)
- b. 皮肤软组织感染(软组织感染、丹毒、甲沟炎、皮肤感染、痈、指(趾)炎)
- c. 局部炎症(鼻窦炎、附睾炎、乳突炎)
- d. 输液相关反应 (输液反应、超敏反应)

- "甲状腺功能检查异常(血促甲状腺激素升高、游离三碘甲状腺原氨酸降低、血促甲状腺激素降低、游离甲状腺素降低、游离甲状腺素升高、甲状腺功能检查异常、游离三碘甲状腺原氨酸升高、三碘甲状腺原氨酸减低、甲状腺素升高、游离三碘甲状腺原氨酸异常、甲状腺球蛋白升高)
- <sup>f</sup> 垂体激素检查异常(血催乳素升高、血促皮质激素减少、血卵泡刺激素增高、血促黄体生成素升高、 血生长激素升高、血促黄体生成素降低、血促皮质激素升高、血卵泡刺激素减低)
  - 8 肾上腺皮质激素检查异常(皮质醇增加、血睾酮降低、皮质醇降低、雌二醇减少、血睾酮升高)
  - h. 食欲下降(食欲下降、消化不良)
  - i. 低蛋白血症(低白蛋白血症、低蛋白血症)
  - j. 失眠 (失眠、睡眠质量差)
  - k. 感觉减退(感觉减退、口腔感觉减退、感觉障碍)
  - 1 肌无力综合征(肌无力、重症肌无力、上睑下垂)
  - m. 外周神经病变 (三叉神经疾病、神经毒性、神经痛)
  - " 心动过速 (窦性心动过速、室上性心动过速、房性心动过速、心动过速、心悸)
- °. 心肌酶谱检查异常(血肌酸磷酸激酶升高、血肌酸磷酸激酶 MB 升高、肌钙蛋白升高、血肌红蛋白升高、肌钙蛋白 T 升高)
  - P. 心律不齐(室性期外收缩、室上性期外收缩、心律不齐、窦性心律不齐、房颤)
  - 9. 肺炎(肺炎、自体免疫性肺部疾病、间质性肺疾病)
  - r. 胸部不适(胸部不适、胸痛)
  - s. 胸腔积液 (胸水、胸腔积液)
  - t. 腹痛 (腹痛、上腹不适)
  - u. 口腔黏膜炎(口腔黏膜炎、嘴唇溃疡形成)
  - v. 消化道出血(胃肠出血、上消化道出血、便血、下消化道出血)
- w. 牙龈牙周疾病(齿龈出血、齿龈肥大、牙疼、牙龈疾病、齿龈疼痛、齿龈炎、牙周炎、牙龈瘤、齿龈肿胀)
  - x. 结直肠炎(结肠炎、直肠炎)
  - y. 功能性胃肠紊乱(功能性胃肠紊乱、胃排空障碍)
  - z. 口咽不适 (口咽不适、咽部炎症)
  - aa. 慢性胃炎 (慢性胃炎、胃炎)
  - bb. 消化道溃疡 (消化道溃疡、胃溃疡)
- <sup>66</sup> 皮疹(皮疹、斑丘疹、带状疱疹、皮疹瘙痒、斑疹、丘疹、皮肤剥脱、脓疱疹、药疹、水疱、血疱、 疱疹病毒感染、脂膜炎)
  - dd. 瘙痒 (瘙痒症、荨麻疹)
  - <sup>ee.</sup> 白癜风(白癜风、色素沉着障碍、皮肤色素减退、皮肤色素脱失)
  - ff. 皮炎(皮炎、痤疮样皮炎、过敏性皮炎、龟头包皮炎)
  - gg. 皮下出血 (瘀点、皮下出血)

- hh. 红斑 (红斑、多形性红斑)
- ii. 肌肉骨骼疼痛(关节痛、背痛、肢体疼痛、肌痛、肌肉骨骼不适、骨痛、肌痉挛、肌肉骨骼疼痛、颈痛、胸部肌肉骨骼疼痛、颌骨疼痛)
  - ji. 关节炎(关节炎、关节病)
  - kk. 肾炎(肾损害、肾病综合征)
  - Ⅱ 水肿 (水肿、眼肿、眼睑浮肿)
  - mm. 疼痛(切口位置疼痛、疼痛、喉部不适、喉部疼痛、口咽疼痛、胸背疼痛)
  - m. 乙型肝炎 DNA 检测阳性 (乙型肝炎 DNA 检测阳性、病毒性肝炎)
- °· 其他实验室检查异常(白细胞增多症、血尿素升高、中性粒细胞增多、总胆汁酸增加、血小板增多症、嗜酸粒细胞增多症、α-羟丁酸脱氢酶升高、单核细胞增多症、降钙素原减少、亮氨酸氨基肽酶升高、脑钠肽激素原增加、血白蛋白升高、血胆红素降低、血免疫球蛋白降低、总蛋白升高、CD8 淋巴细胞百分率增高、C反应蛋白升高、T-淋巴细胞计数升高、平均细胞血红蛋白降低、平均细胞血红蛋白浓度降低、嗜碱性粒细胞增多症、嗜酸粒细胞减少症、血胆碱酯酶降低、血胆碱酯酶升高、血葡萄糖降低)
- PP 凝血功能检查异常(活化部分凝血活酶时间延长、凝血酶原时间延长、纤维蛋白 D-二聚体升高、凝血试验异常、血纤维蛋白原降低、抗凝血酶Ⅲ抗体减少、纤维蛋白降解物升高、血纤维蛋白原升高)
- 49· 其他电解质紊乱(低氯血症、低镁血症、高钙血症、高钾血症、血铁降低、低钙血症、高镁血症、电解质失调、高氯血症、高钠血症、血钙降低、血钙升高)
- ". 其他尿常规检查异常(尿中尿胆原增加、尿白细胞阳性、色素尿、尿胆红素升高、尿晶体检出、尿糖检出、尿酮体存在、尿比重升高、尿亚硝酸盐检出)
- ss. 其他心电图检查异常(心电图 T 波异常、起搏点游走、心电图 ST 段异常、心电图 ST-T 段异常、心电图 T 波波幅降低、右束支阻滞、QRS 轴异常、心电图示低电压)

#### 【注意事项】

反应性毛细血管增生症

反应性毛细血管增生症,大多发生在体表皮肤,少数可见于口腔黏膜、鼻腔黏膜 以及眼睑结膜。发生于皮肤的反应性毛细血管增生,初始多表现为体表鲜红色点状 物,直径≤2 mm,随着用药次数增加,病变范围可逐渐增大,多为结节状,也有斑 片状,颜色鲜红或暗红,需观察临床症状和体征,可参照以下分级标准和治疗建议 进行处理:

| 分级† | 临床表现 | 治疗建议 |
|---|---|---|
| 1级 | 单个最大直径<br>≤10 mm,伴或不伴破<br>溃出血 | 继续用药,易摩擦部位可用纱布保护,避免出血。破溃出血者可采用局部压迫止血治疗。 |
| 2级 | 单个最大直径>10 mm,<br>伴或不伴破溃出血 | 继续用药,易摩擦部位可用纱布保护,<br>避免出血。破溃出血者可局部压迫止血,<br>或采取局部治疗措施,如激光或手术切 |

| | | 除等。避免破溃处感染。 |
|---|---|---|
| 3级 | 呈泛发性,可以并发皮<br>肤感染,可能需要住院<br>治疗 | 暂停用药,待恢复至≤1级后恢复给药,<br>易摩擦部位可用纱布保护,避免出血。<br>破溃出血者可局部压迫止血,或采取局<br>部治疗措施如激光或手术切除等,并发<br>感染者给予抗感染治疗。 |
| 4级‡ | 多发和泛发,威胁生命 | 永久停药 |
| 5级‡ | 死亡 | |

†分级依据《CSCO 免疫检查点抑制剂相关的毒性管理指南 2019》。

‡卡瑞利珠单抗研究中未发生4级危及生命和5级死亡不良事件。

当患者出现该不良反应时,应避免抓挠或摩擦,易摩擦部位可用纱布保护以避免 出血,同时应联系医生,获得恰当的处理建议。破溃出血者可采用局部压迫止血, 反复出现者可于止血后于皮肤科就诊,采取如激光或手术切除等局部治疗。局部并 发感染者应给予局部抗感染治疗。反应性毛细血管增生症可能在皮肤以外的其他组 织发生(包括睑结膜、内外眦、口腔黏膜、咽喉等消化道黏膜或其它脏器),应根 据自查体征和症状,必要时就医进行相应医学检查,如大便潜血、内窥镜及影像学 检查(具体相关内容详见《反应性毛细血管增生症信息收集及风险管理计划》)。

更多不良反应数据详见卡瑞利珠单抗说明书。

### (3) 化疗引起的不良反应如下:

#### a) 奥沙利铂

胃肠道反应:腹泻、恶心、呕吐以及粘膜炎、腹痛、便秘,消化不良、胃食道反流、 胃肠道出血,肠梗阻、结肠炎;

血液系统:白细胞、中性粒细胞减少;血小板、出血及凝血异常:出血、血尿、深静脉血栓、直肠出血、血栓栓塞事件、贫血;

心血管系统: 高血压;

神经系统反应:常见的过敏反应包括支气管痉挛、血管性水肿、低血压、胸痛感以及过敏性休克。出现外周感觉神经病变,包括头痛、感觉异常、味觉异常,急性神经感觉症状,运动神经炎、构音障碍;

肾脏以及泌尿系统异常:排尿困难、尿频和排尿异常,蛋白尿,血尿素氮和肌酐水平升高;

生化异常: 轻中度转氨酶和碱性磷酸酶水平升高、胆红素升高、血糖异常、LDH 升高、低钾血症、低白蛋白血症。

更多不良反应数据详见奥沙利铂说明书。

b) 氟尿嘧啶

恶心、食欲减退或呕吐,一般剂量多不严重;

偶见口腔粘膜炎或溃疡,腹部不适或腹泻;

外周血白细胞减少常见,大多在疗程开始后 2-3 周内达到最低点,约在 3-4 周内恢复 正常,血小板减少罕见:

极少见咳嗽、气急或小脑共济失调:

脱发或注入药物的静脉上升性色素沉着:

静脉滴注处药物外溢可引起局部疼痛、坏死或蜂窝组织炎;

长期应用可致神经系统毒性;

偶见用药后心肌缺血, 可出现心绞痛和心电图变化。

更多不良反应数据详见氟尿嘧啶说明书。

(4) 采血/活检的风险: 采血的部位可能会出现疼痛或者淤血。您也可能感觉到眩晕。 采血的部位也有可能出现感染。如果您需要进行活检以获得肿瘤组织,活检的部位 可能会出现疼痛,不适或者瘀血。在少数情况下也可能出现和手术相关的并发症, 例如感染,出血等以及与活检部位相关的并发症。

如出现相关的常见不良反应,负责您的医生将会观察、检查及随访您的情况,根据您的情况给予相应的治疗。毒副反应将严格记录在病例报告表中,判断其性质、严重程度以及评估与试验的相关性。希望您在参与研究过程中遵循医嘱,积极配合治疗,按照试验方案的要求接受观察和随访,需要您提前合理安排。

(4) 如您正处于怀孕期或在研究期间受孕,该研究干预措施或治疗可能对胚胎或胎 儿造成目前无法预知的风险。

#### 【研究治疗结束/提前终止研究治疗】

受试者出现以下的任何一种情况,必须停止治疗,但可继续在研究中接受监测:

- 1. 影像学证据表明肿瘤进展;
- 2. 受试者撤回知情同意,要求退出研究;

- 3. 无法耐受毒性者;
- 4. 受试者依从性不佳;
- 5. 受试者失访;
- 6. 研究者认为有必要退出研究的情况。

### 【受试者的医疗处理】

在临床试验和随访期间,对于受试者出现与试验相关的不良事件,包括有临床意义的 实验室异常时,研究者和临床试验机构应当保证受试者得到妥善的医疗处理,并将相关情况 如实告知受试者。研究者意识到受试者存在合并疾病需要治疗时,应当告知受试者,并关注 可能干扰临床试验结果或者受试者安全的合并用药。

#### 【研究获益】

参加该临床研究将获得免费索凡替尼与卡瑞利珠单抗免费赠药,直至退组,同时卡瑞利珠单抗最多用药两年,化疗用药及其他药物以及检查费用需要您自费。

### 【受试者隐私保护】

如果您决定参加本项研究,您参加研究及在研究中的个人资料均属保密。您的血标本或组织标本将以研究编号数字而非您的姓名加以标识,检验中心为中山大学附属肿瘤医院,您就诊检查所产生的医疗废弃物按照中心常规医疗废物处置管理制度执行清理。您的生物标本将仅用于科研探索,研究者将确保您的样本信息安全。您的身份不会被识别,可以识别您身份的信息将不会透露给研究小组以外的成员,除非获得您的许可。所有的研究成员都被要求对您的身份保密。您的档案将保存在有锁的档案柜中,仅供研究人员查阅。为确保研究按照规定进行,必要时,政府管理部门或伦理审查委员会的成员按规定可以在研究单位查阅您的个人资料。这项研究结果发表时,将不会披露您个人的任何资料。

#### 【其他医疗方案】

您目前的疾病状态的标准治疗推荐体能状态良好的患者接受纳米脂质体伊利替康联合5-FU/LV,其他推荐方案还包括:一线使用吉西他滨为基础的方案,二线建议以5-FU 为基础的方案;一线使用5-FU 类为基础的方案,二线建议使用吉西他滨为基础的方案;对于术后发生远处转移者,若距离辅助治疗结束时间>6 个月,除选择原方案全身化疗外,也可选择替代性化疗方案或者参加临床研究。本研究在标准治疗的基础上联合抗血管生成药物以及免疫治疗以期待进一步提高疗效。除了参加本研究,请您和您的医生讨论其它可选的医疗方

案,例如化疗药物、其他靶向药物、免疫治疗等治疗手段。您的研究医生会与您讨论可能的 风险以及其它治疗方法的优劣。请您在与医生充分讨论其他可能采取的方案后,再决定是否 参加本研究。

### 【潜在获益】

如果您同意参加本研究,从您的治疗经过中得到的数据将使医生能更好地治疗像您那样的病人,这对未来的患者很有帮助。

您的肿瘤可能得到控制并进行手术治疗,生存可能延长。然而,和大多数的治疗一样,本研究的治疗也可能不能控制您的疾病。

# 【受试者伤害赔偿】

如果由于参加本临床研究,在您遵从研究医生指令行事的前提下,发生了与研究相关的 伤害,您将获得必要的医疗治疗。对发生与试验相关的损害或死亡,将按中国的法律法规获 得赔偿。

### 【退出研究】

您可以选择不参加本项研究,或者在任何时候通知研究者要求退出研究,您的数据将不纳入研究结果,您的任何医疗待遇与权益不会因此而受到影响。

如果您需要其它治疗,或者您没有遵守研究计划,或者发生了与研究相关的损伤或者有 任何其它原因,研究医师可以终止您继续参与本项研究。告知受试者可能被终止试验的情况 以及理由。

#### 【联系】

您可随时了解与本研究有关的信息资料和研究进展,如果您有与本研究有关的问题,或您在研究过程中发生了任何不适与损伤,或有关于本项研究参加者权益方面的问题您可以通过\_\_\_\_\_(<u>电话号码</u>)与\_\_\_\_\_(<u>研究者或有关人员姓名</u>)联系。

如果在研究过程中您有关于伦理方面的问题,可以联系中山大学肿瘤防治中心伦理委员会:联系电话: 020-87343009。

# 知情同意书

我已经阅读了本知情同意书。

我有机会提问而且所有问题均已得到解答。

我理解参加本项研究是自愿的。

我的个人身份信息将会被保密。

我可以选择不参加本项研究,或者在任何时候通知研究者后退出,我的任何医疗待遇与权益不会因此而受到影响。

如果我需要其它治疗,或者我没有遵守研究计划,或者发生了与研究相关的损伤或者有任何其它原因,研究医师可以终止我继续参与本项研究。

我将收到一份签过字的"知情同意书"副本。

| | 受试者姓名: | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | 受试者签名: | | | | - | | | |
| | 日期: | 年 | _月 | 目 | | | | |
| | 我已准确地将 | 这份文本告知 | 印受试者, | 他/她 | 准确地阅 | ]读了这份 | 知情同意书 | ,受试者有机 |
| 会提 | 出问题。 | | | | | | | |
| | 研究者姓名: | | | | | | | |
| | 研究者签名: | | | | - | | | |
| | 日期: | 年 | _月 | 目 | | | | |
| | (注, 加果受 | 试者无行为的 | 能力时则多 | <i>雪洋完/</i> | <b>半理 / 冬</b> | 夕) | | |